CLINICAL TRIAL: NCT01248936
Title: A SINGLE ARM, OPEN LABEL, EXPANDED ACCESS STUDY OF RG7204 IN PREVIOUSLY TREATED PATIENTS WITH METASTATIC MELANOMA
Brief Title: A Study of RO5185426 in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25597
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Overall Trial (Experimental): Participants received vemurafenib 960 milligram (mg) orally two times a day for up to one year. Participants were treated until disease progression, unmanageable toxicity most probably attributable to vemurafenib, withdrawal of consent, and study termination by the sponsor
  Interventions: Drug: RO5185426

INTERVENTIONS:
Drug: RO5185426

SUMMARY:
This is an open-label, non-comparative, multicenter, expanded access study of RO5185426 in patients who have received prior systemic therapy for metastatic melanoma and who have no other satisfactory treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic melanoma with documented BRAF V600E mutation, determined by the cobas BRAF V600 mutation test
* Patients with either measurable or non-measurable disease
* Adequate recovery from most recent systemic or local treatment for metastatic melanoma
* Adequate organ function
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of RO5185426
* For men with female partners of childbearing potential, agreement to use a latex condom, and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of RO5185426
* Negative serum or urine pregnancy test within 7 days of commencement of treatment in premenopausal women. Women who are either surgically sterile or have been post-menopausal for at least 1 year are eligible to participate in this study
* Agreement not to donate blood or blood products during the study and for at least 6 months after discontinuation of RO5185426; for male patients, agreement not to donate sperm during the study and for at least 6 months after discontinuation of RO5185426

Exclusion Criteria:

* Pregnant or breast-feeding
* Concurrent anti-tumor therapy
* Uncontrolled medical illness
* History of congenital prolonged QT syndrome or patients with a mean QTc interval greater than 470 milliseconds at baseline, or ongoing grade 2 or greater cardiac arrhythmia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (23):
  - Tucson, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Santa Monica, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Palm Harbor, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Park Ridge, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - New York, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
  - Seattle, Washington

REFERENCES:
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 29 study sites in the United States (US). The study period was from 10 December 2010 to 24 October 2011.
Pre-assignment Details: Overall, 745 participants were screened during the study, of which 374 were enrolled to receive study treatment; the main reason for screen failure was negative cobas test, consent withdrawal, BRAF test not performed, patient died or progressed, and other unspecified reasons. Of 374 participants, 3 did not receive treatment after enrollment.
Period: Overall Study
Arm/Group | Overall Trial
Started | 374
Completed | 0
Not Completed | 374
Not completed — Sponsor Decision | 259
Not completed — Progression of Disease | 50
Not completed — Death | 26
Not completed — Withdrawal of Consent | 20
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 7
Not completed — Refused Treatment | 1
Not completed — Other reason | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received at least one dose, or a partial dose of vemurafenib. Three participants who were enrolled did not receive vemurafenib hence not included in safety population.
Groups:
- Overall Trial: Participants received vemurafenib 960 mg orally two times a day for up to one year. Participants were treated until disease progression, unmanageable toxicity most probably attributable to vemurafenib, withdrawal of consent, and study termination by the sponsor.
Arm/Group | Overall Trial
Number analyzed (Participants) | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (13.8)
Age, Customized [Number; unit: participants]
  Adolescents (12-17 year) | 1
  From 18 - 64 years | 289
  From 65 - 84 years | 79
  Over 85 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 229

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Best Overall Response (Unconfirmed)
Description: The best overall response (unconfirmed) is the best response recorded from the start of the treatment until disease progression/recurrence which was unconfirmed. Participants were assessed for best overall response by investigator as per 'Response Evaluation Criteria in Solid Tumors' (RECIST v1.1).
Time Frame: Up to 1 year
Population: The efficacy population was defined as treated participants who had measurable disease at baseline and at least one post-baseline tumor assessment.
Measure: Number; unit: participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 241
participants | 129

2. Secondary Outcome: Number of Participants With Best Overall Response (Unconfirmed) by ECOG Performance
Description: The best overall response recorded from the start of the treatment until disease progression/recurrence which was unconfirmed in patients with Eastern Cooperative Oncology Group (ECOG) performance status 2 or 3/0 or 1. Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair. 5: Dead. This endpoint was tumor response category according to investigator assessment per RECIST v1.1 for efficacy assessment. The 'n' is number of participants with ECOG performance status in each criteria.
Time Frame: Up to 1 year
Population: The efficacy population was defined as treated patients who had measurable disease at baseline and at least one post-baseline tumor assessment.
Measure: Number; unit: Participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 241
Participants
  ECOG performance status 2 or 3; n=31 | 13
  ECOG performance status 0 or 1; n=210 | 116

3. Secondary Outcome: Number of Participants With Best Overall Response (Confirmed)
Description: The best overall response (confirmed) is the best response recorded from the start of the treatment until disease progression/recurrence which was confirmed. Participants were assessed for best overall response by investigator as per RECIST v1.1.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 241
Participants | 26

4. Secondary Outcome: Number of Participants With Best Overall Response (Confirmed) by ECOG Performance
Description: The best overall response recorded from the start of the treatment until disease progression/recurrence which was confirmed in patients with Eastern Cooperative Oncology Group (ECOG) performance status 2 or 3/0 or 1. Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair. 5: Dead. Participants were assessed for best overall response by investigator as per RECIST v1.1. The 'n' is number of participants with ECOG performance status in each criteria.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 241
Participants
  ECOG performance status 2 or 3); n= 31 | 1
  ECOG performance status 0 or 1); n= 210 | 25

5. Secondary Outcome: Mean Time to Complete Response/Partial Response
Description: Mean time to Complete Response (CR)/Partial Response(PR) (confirmed or unconfirmed was assessed). Participants were assessed for best overall response by investigator as per RECIST v1.1.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Overall Trial
Number analyzed (Participants) | 241
Months
  Mean time to confirmed CR or PR | 1.8 (0.3)
  Mean time to unconfirmed CR or PR | 2.0 (0.7)

6. Primary Outcome: Number of Participants With Any Adverse Event, Adverse Events With Severity, Adverse Events Leading to Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs will be graded according to the 'National Cancer Institute Common Terminology Criteria for Adverse Events' (NCI CTCAE, v4.0). However Laboratory data will be summarized by grade using the NCI CTCAE, v4.0 toxicity grade.
Time Frame: Up to 1 year
Population: The safety population was defined as participants who received at least one dose, or a partial dose, of vemurafenib.
Measure: Number; unit: participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 371
participants
  Any AE | 346
  Grade 3 AEs | 115
  Grade 4 AEs | 15
  Grade 5 AEs | 7
  AEs leading to discontinuation | 9

7. Primary Outcome: Number of Participants With Any Serious Adverse Event, Death and Cause of Death
Description: Serious Adverse Event (SAEs) is defined as those events that were fatal or immediately life-threatening, and those events that resulted in hospitalization; prolonged an existing hospitalization; resulted in disability; or was a congenital anomaly. Number of participants who died and the cause of death are also recorded.
Time Frame: Up to 1 year
Population: The safety population was defined as participants who received at least one dose, or a partial dose, of vemurafenib.
Measure: Number; unit: participants
Arm/Group | Overall Trial
Number analyzed (Participants) | 371
participants
  Any SAEs | 83
  All Deaths | 43
  Death due to progression of disease | 22
  Death due to adverse event | 8
  Deaths which are not related to study drug | 6
  Deaths which are related to study drug | 2

ADVERSE EVENTS:
Time Frame: Up to 1 Year
Description: Serious adverse events and non-serious adverse events are reported in safety analysis set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | Overall Trial
Serious Adverse Events (participants affected / at risk) | 83/371
Other Adverse Events (participants affected / at risk) | 308/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Trial (N=371)
Vomiting (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diverticular Perforation (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Bacterial Infection (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pyrexia (General disorders) | 5
Death (General disorders) | 2
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Drug Withdrawal Syndrome (General disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 1
Convulsion (Nervous system disorders) | 5
Headache (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Lumbar Radiculopathy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Failure To Thrive (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Electrocardiogram Qt Prolonged (Investigations) | 3
Blood Bilirubin Increased (Investigations) | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1
Blood Uric Acid Increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 3
Mental Status Changes (Psychiatric disorders) | 2
Paranoia (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Renal Colic (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Pupils unequal (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Trial (N=371)
Rash (Skin and subcutaneous tissue disorders) | 102
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 62
Alopecia (Skin and subcutaneous tissue disorders) | 41
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 29
Dry Skin (Skin and subcutaneous tissue disorders) | 26
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 23
Pruritus (Skin and subcutaneous tissue disorders) | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 136
Myalgia (Musculoskeletal and connective tissue disorders) | 30
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 20
Fatigue (General disorders) | 102
Oedema Peripheral (General disorders) | 41
Pyrexia (General disorders) | 37
Nausea (Gastrointestinal disorders) | 69
Diarrhoea (Gastrointestinal disorders) | 42
Vomiting (Gastrointestinal disorders) | 30
Constipation (Gastrointestinal disorders) | 20
Sunburn (Injury, poisoning and procedural complications) | 48
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23
Decreased Appetite (Metabolism and nutrition disorders) | 42
Headache (Nervous system disorders) | 37
Weight decreased (Investigations) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.